CLINICAL TRIAL: NCT07376603
Title: Intensity-Modulated Radiotherapy Alone for Stage IB Nasopharyngeal Carcinoma Without High-Risk Features
Brief Title: IMRT Alone for Stage IB Nasopharyngeal Carcinoma Without High-Risk Features
Status: Recruiting | Type: Observational
Sponsor: Qiaojuan Guo (Other Government)
Responsible Party: Sponsor-Investigator, Qiaojuan Guo, Professor, Fujian Cancer Hospital
Organization: Fujian Cancer Hospital (Other Government)
Other Study IDs: NPC0013.1
Record Dates: First submitted 2026-01-17; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Intensity-modulated Radiotherapy; Stage IB
Keywords: Nasopharyngeal Cancinomar; Stage IB; RT along

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IMRT along: IMRT Alone for 169 Patients with Stage IB Nasopharyngeal Carcinoma Without High-Risk Features
  Interventions: Radiation: IMRT along

INTERVENTIONS:
Radiation: IMRT along — All patients administered with definitive radiotherapy

SUMMARY:
This observational study aims to evaluate the efficacy and safety of intensity-modulated radiotherapy (IMRT) alone in patients with stage IB nasopharyngeal carcinoma (NPC) without high-risk features. The primary objective is to determine the therapeutic effectiveness of this approach

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed, newly diagnosed nasopharyngeal carcinoma 3. Age 18-70 years 4. Stage IB disease (T1-2N1M0) per the 9th edition AJCC/UICC staging system 5. Upper-neck nodal metastasis only: inferior border of every positive node at or above the inferior border of the hyoid bone 6. ECOG performance status 0-2 7. Adequate bone-marrow function

Exclusion Criteria:

1. Age > 70 years or < 18 years
2. Matted lymph nodes: two or more contiguous nodes with loss of intervening fat planes and/or extracapsular extension forming a confluent mass
3. Largest metastatic lymph-node ≥ 3 cm in the longest dimension
4. Lower-neck nodal metastasis: inferior border of any positive node below the inferior border of the hyoid bone
5. Prior malignancy except adequately treated basal-cell or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix
6. Pregnancy or lactation (serum pregnancy test required for women of child-bearing potential; effective contraception mandatory during treatment)
7. Previous radiotherapy to the head-and-neck region
8. Prior chemotherapy or surgery for the primary tumour or metastatic nodes (diagnostic procedures excluded)
9. Any severe comorbidity that would confer unacceptable risk or compromise protocol adherence, including but not limited to unstable cardiac disease, renal failure, chronic hepatitis, or uncontrolled psychiatric disorder
10. History of severe hypersensitivity reactions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IB NPC
Sampling Method: Non-Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival | 3-year
  Time from diagnosis to the disease relapse (either locoregional recurrence or distant metastasis) or death from any cause.

SECONDARY OUTCOMES:
Locoregional Relapse-Free Survival | 3-year
  Time from diagnosis to first documented locoregional recurrence before the last follow-up visit.
Distant Metastasis-Free Survival | 3-year
  Time from diagnosis to first documented distant metastasis before the last follow-up visit
Overall Survival | 3-year
  Time from diagnosis to death from any cause or to the last follow-up visit for patients still alive.
Safety of Radiation | at inclusion, 3 months, 6 months,12 months, 24 months, 36 months, and 60 months
  Acute and late radiation toxicities were graded with the CTCAE criteria
Quality of life (EORTC QLQ C30) | at inclusion, 3 months, 6 months,12 months, 24 months, 36 months, and 60 months.
  Quality of life score was calculated according to the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ C30), the range is 0-100, higher scores mean a worse outcome.
Quality of life score QLQ-HN35 | at inclusion, 3 months, 6 months,12 months, 24 months, 36 months, and 60 months.
  The quality of life score was calculated according to the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire QLQ-HN35; the range is 0-100, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol